CLINICAL TRIAL: NCT03749161
Title: Comparison Between Bilateral Low-add Multifocal Intraocular Lenses and Monofocal Intraocular Lenses: A Randomised Trial
Brief Title: Low-add Multifocal vs. Monofocal IOLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oculentis
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract Surgery; Low-add intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lentis comfort (Experimental): Patient will receive the low-add multifocal IOL during cataract surgery
  Interventions: Device: Low-add multifocal IOL
- Lentis L-313 (Experimental): Patient will receive the monofocal IOL Lentis L-313 during cataract surgery
  Interventions: Device: Monofocal IOL

INTERVENTIONS:
Device: Low-add multifocal IOL — Lentis comfort, low-add multifocal, IOL
  Arms: Lentis comfort
Device: Monofocal IOL — Lentis L-313, monofocal IOL
  Arms: Lentis L-313

SUMMARY:
Compare low-add multifocal IOLs with monofocal IOLs to evaluate if patients in the low-add multifocal IOL group have better unaided distance visual acuity compared to the monofocal group.

DETAILED DESCRIPTION:
Spectacle independence is one of the main aims in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia or low myopia, leads to high levels of patient satisfaction in distance vision, spectacle dependence for intermediate vision, reading and other near vision tasks is the usual result.

There are different techniques to reduce spectacle dependence, the most common one is the use of multifocal IOLs. However, a variable number of patients complain of problems, such as glare or haloes (positive dysphotopsia symptoms). Dysphotopsia symptoms may vary significantly from patient to patient. The real incidence of dysphotopsia like symptoms after cataract surgery and multifocal IOL is unknown and the implantation of multifocal IOLs is a commonly accepted contraindication in patients who are night drivers. Another characteristic of many multifocal IOLs is that it can provide patients with excellent near and distance vision but lack in the intermediate range.

One option to enhance intermediate vision and to leave patients with good contrast sensitivity is the use of low-add multifocal IOLs. These IOLs are adequate to expectations a lot of patients have, who were used to have a good distance vision and who were wearing spectacles when performing near vision tasks before surgery. Many of these patients would prefer to keep their reading spectacles after surgery and ideally would like to function well at distance and intermediate (60 to 80 cm - computer distance, household work…) range without glasses.

One example of these low-add multifocal IOLs is the LENTIS Comfort MF15 with a near add of 1.50D (on IOL plane). Its single, blended transition zone works to deliver patients the same kind of distance vision as a monofocal IOL with the addition of enhanced intermediate vision. In particular, this design provides improved vision at a distance of 60 cm and more. Additional key features of the Comfort IOL include good contrast sensitivity for twilight vision, optimized depth of focus, and natural imaging quality and color sensitivity. Especially this type of IOL may lead to more tolerance of postoperative refractive errors due to biometry and IOL power calculation imprecision. This should result in better unaided distance vision and therefore higher patient satisfaction after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract in both eyes
* Scheduled for bilateral cataract surgery
* Motivated to be less spectacle dependant in the distance to intermediate vision range
* Patients with an expected BCDVA of 0.8 snellen score or better after surgery
* Patients with the need of an IOL Power in the range of 10 to 30D (biometry performed with the IOL master 700)
* Age 21 and older
* Written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Retinopathia pigmentosa
* Chronic uveitis
* Amblyopia
* Pupil decentration > 1mm center shift
* preceded retinal surgery
* preceded Laser-in-situ-Keratomileusis (LASIK)
* Any ophthalmic abnormality that could compromise visual function or the measurements

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Spectacle independence questionnaire | 12 months
  Spectacle independence will be assessed using a questionnaire. In this questionnaire the patient will be asked about usage of spectacles for far, near and intermediate distance. Best result will be if the patient is independent from any spectacles in the different distances.

SECONDARY OUTCOMES:
Best Corrected Distance Visual Acuity and Uncorrected Intermediate Visual Acuity | 12 months
  Best corrected distance and uncorrected intermediate visual acuity will be assessed using the ETDRS charts
Titmus Fly Stereo test | 12 months
  Stereo Vision assessment will be done using the Titmus Fly Stereo test. The patients will be asked to detect stereoscopic objects of different difficulty levels. The result will be better, the more correct stereoscopic objects the patient will detect.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided